CLINICAL TRIAL: NCT04342481
Title: To Explore the Educational Experience of UK Primary Care Health Practitioners for Peripheral Arterial Disease (PAD), Including Identification of Factors That Shape Their Preferred Learning Style and Assess Health Professionals Opinions of PAD Recognition and Management
Brief Title: Education and Management of PAD in Primary Care
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); The George Davies Charitable Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0782/280635
Record Dates: First submitted 2020-04-08; First posted 2020-04-13 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2021-09

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; peripheral artery disease; PAD - peripheral arterial disease; PAD
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Educational Screening tool — Educational Screening tool

SUMMARY:
Peripheral arterial disease (PAD) occurs when the vessels carrying blood to the legs become narrowed or blocked. It affects 1 in 5 people aged over 60 and are at risk of losing their leg, developing a heart attack or stroke, or die early.

Early symptoms of peripheral arterial disease (PAD) include aching in the legs when walking which may not be recognised by healthcare professional. Our research has shown that knowledge and recognition of PAD is poor in healthcare professionals and trainees. There appears to be little time provided within healthcare professional training for PAD.

To improve PAD recognition/management, the investigators want to identify the current level of training given to healthcare professionals; opinion towards PAD related to their training and how they prefer to receive training.

With the information gained from this research, the development of an educational training package for GPs, practice nurses and their trainees to improve recognition of PAD is anticipated.

DETAILED DESCRIPTION:
Around 20% of people above 60 years are estimated to have PAD. The prevalence of PAD is expected to rise due to a sedentary life-style, poor dietary choices, rising prevalence of diabetes and longer life-expectancy.

The most common presentation of symptomatic PAD is intermittent claudication - pain on activity. In some cases the reduction in blood flow is so severe that it causes pain at rest, ulceration or gangrene (chronic limb threatening ischemia, CLTI). Approximately 5% of individuals between the age of 55 and 74 in the UK have IC or CLTI. Compared to age-matched individuals, these patients are more likely to suffer cardiovascular events - heart attack and strokes and cognitive impairment (10). Of those with IC, 5% will progress to CLTI. In patients with CLTI the one-year risk of limb amputation is 30% and five-year all-cause mortality is 50%, similar to various advanced forms of cancer. Recognition and management are essential to reducing the limb and life loss sequela.

Management of these high-risk individuals is shared between primary care (diagnosis, treatment of cardiovascular risk-factors, rehabilitation) and secondary care (vascular reconstruction, amputation, specialist management of cardiovascular disease).

This mutli-centre prospective cohort study will investigate the explore the educational experience of UK primary care health practitioners for peripheral arterial disease (PAD), including identification of factors that shape their preferred learning style and assess health professionals opinions of PAD recognition and management.

ELIGIBILITY:
Inclusion Criteria:

1. Practising healthcare practitioners within primary care
2. Participants must be aged 18 years or older
3. Participants must be able to access the online questionnaire
4. Participants must have the capacity to consent
5. Participants should speak English

Exclusion Criteria:

1. Healthcare practitioners who are not in practice.
2. Participants who do not consent
3. Participants who are unable to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Practising healthcare practitioners within primary care
Sampling Method: Probability Sample
Enrollment: 891 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Educational exposure do primary care health practitioners experience regarding PAD | 10 years
  Educational exposure do primary care health practitioners experience regarding PAD

SECONDARY OUTCOMES:
What opinions do UK primary care health practitioners have towards PAD recognition and management? | 10 years
  What opinions do UK primary care health practitioners have towards PAD recognition and management?

OTHER OUTCOMES:
What factors are important when considering educational interventions to healthcare practitioners in primary care? | 10 years
  What factors are important when considering educational interventions to healthcare practitioners in primary care?

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leicester, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised dataset will be available on request to the Chief Investigator (Prof Rob Sayers).